CLINICAL TRIAL: NCT06379503
Title: Effect of Heart Yoga Applıed To Patıents Undergoıng Cardıovascular Surgery on Sleep, Depressıon And Qualıty of Lıfe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Kubra Oymaagaclio, specialist nurse, Dokuz Eylul University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021/37-04
Record Dates: First submitted 2024-04-03; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Disease; Yoga; Nursing Caries
Keywords: Yoga; Heart Surgery; Nursing
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Heart yoga practice for 12 weeks on 30 patients who underwent heart surgery
  Interventions: Other: HEART YOGA
- control (Active Comparator): routine nursing care
  Interventions: Other: routine nursing care

INTERVENTIONS:
Other: HEART YOGA — Heart yoga; It includes regular, balanced, safe light physical exercises, breathing exercises that provide breathing control, and meditation practices that include relaxation techniques.
  Arms: intervention
Other: routine nursing care — Basic nursing care after heart surgery
  Arms: control

SUMMARY:
This type of study is a randomized controlled trial. The aim is to contribute to the literature by comparing the effects of heart yoga on the depression level, sleep and quality of life of patients who do and do not do heart yoga.

The main elements it aims to answer are:

* Heart yoga applied to patients who have undergone heart surgery improves their sleep quality compared to those who have not.
* Heart yoga applied to patients who have undergone heart surgery reduces the level of depression compared to those who have not.
* Heart yoga applied to patients who have undergone heart surgery increases the quality of life compared to those who have not.

Patients who accept the study will practice heart yoga simultaneously with heart yoga videos via an online link every other day for 12 weeks after heart surgery.

Researchers will compare intervention and control groups to see if there are any effects on sleep quality, depression level, and quality of life.

DETAILED DESCRIPTION:
In order to collect the data of the study, Personal Information Form, Physiological Parameters, Pittsburgh Sleep Quality Index (PUKI), Beck Depression Inventory, World Health Organization Quality of Life Scale-Short Form were used to evaluate the individual characteristics of the patient and were collected from patients who underwent cardiovascular surgery. (Permission to use scale has been obtained.) The researcher received a certificate by participating in a national and international certified training program of 200 hours of basic yoga and 250 hours of yoga therapy training. The "Heart Yoga Guidance Booklet" was developed by the researcher in line with the guide prepared for the practice of heart yoga, the training received, literature reviews on the subject and clinical experiences. In line with this booklet, videos were created for patients to apply at home. It was easily accessible by providing an online link. In addition, a monitoring form was given every other day to ensure controlled follow-up of the patients.

The patients were randomized and the study started with patients who accepted the study. The suitability and clarity of the scales were checked with pre-application (n: 20).

In addition to routine nursing care, patients in the intervention group received heart yoga every other day for 70-80 minutes a day, starting from the 1st postoperative week until the end of the 12th week. The control group continued routine nursing care.

Evaluation scales were filled in by the patients before surgery, at the 1st week after surgery, at the 1st month after surgery, and finally at the 3rd month after surgery.

ELIGIBILITY:
Research Inclusion Criteria

* Those who have undergone cardiovascular surgery,
* Those who are over 18 years old,
* Oriented to person, place and time,
* Extubated on the first day after surgery,
* Pain control was achieved before the application,
* Those who do not practice yoga or similar practices,
* No verbal communication disability (hearing and speaking),
* No physical mobility problems,
* No obstacle to using technology,
* Patients who volunteered to participate in the study were included in the study. Exclusion Criteria
* Having low blood pressure,
* The amount of drainage from the chest tube is excessive, which hinders cardiac yoga movements,
* Those who have conditions such as asthma, chronic obstructive pulmonary disease (COPD),
* Patients with diagnosed psychiatric and neurological disorders were excluded from the study.

Criteria for Exclusion from the Study

* Unable to communicate during the research process,
* Patients who wanted to leave the study during the research period were excluded from the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
sleep quality | 12 week
  Pittsburgh Sleep Quality Index (PSQI)
depression | 12 week
  Beck Depression Inventory (BDI)
life quality | 12 week
  World Health Organization Quality of Life Scale (WHOQOL - BREF)

CONTACTS AND LOCATIONS:
Overall Officials: Sonay Göktaş, Prof. dr., Principal Investigator — Sağlık Bilimleri Universty
Locations (1):
- Dokuz Eylül Üniversitesi Hastanesi, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emoto T, Yamashita T, Sasaki N, Hirota Y, Hayashi T, So A, Kasahara K, Yodoi K, Matsumoto T, Mizoguchi T, Ogawa W, Hirata K. Analysis of Gut Microbiota in Coronary Artery Disease Patients: a Possible Link between Gut Microbiota and Coronary Artery Disease. J Atheroscler Thromb. 2016 Aug 1;23(8):908-21. doi: 10.5551/jat.32672. Epub 2016 Mar 5. PMID 26947598
- [Background] Ball L, Costantino F, Pelosi P. Postoperative complications of patients undergoing cardiac surgery. Curr Opin Crit Care. 2016 Aug;22(4):386-92. doi: 10.1097/MCC.0000000000000319. PMID 27309972
- [Background] Chrastina J, Novak Z, Brichta J, Pavlik P, Riha I, Nemec P. Neurosurgical treatment of cerebrovascular complications of heart surgeries and interventions. Turk Neurosurg. 2014;24(6):897-905. doi: 10.5137/1019-5149.JTN.10240-13.0. PMID 25448207
- [Background] Smeltzer, S. C., Bare, B.G., Hinkle, J. L., Cheever, K. H. (2010). Postoperative Nursing Management. In: Brunner & Suddarth's Textbook of Medical-Surgical Nursing, 12th.ed. China: Wolters Kluwers Health/Lippincott Williams&Wilkins; 461-478.
- [Background] Shafiq A, Jayaram N, Gosch KL, Spertus JA, Buchanan DM, Decker C, Kosiborod M, Arnold SV. The Association Between Complementary and Alternative Medicine and Health Status Following Acute Myocardial Infarction. Clin Cardiol. 2016 Aug;39(8):440-5. doi: 10.1002/clc.22559. Epub 2016 May 31. PMID 27244586
- [Background] Erdoğan Z, Oğuz S, Erol E. (2012). Use of complementary therapies in the patients with heart disease. Spatula DD; 2(3):135-9.
- [Background] Haefner J. Complementary and Integrative Health Practices for Depression. J Psychosoc Nurs Ment Health Serv. 2017 Dec 1;55(12):22-33. doi: 10.3928/02793695-20170905-02. Epub 2017 Sep 12. PMID 28892554
- [Background] Şahin N, Aydın D, Akay B. (2019). The attitudes of nursing students towards holistic complementary and alternative medicine. Balıkesir Health Sciences Journal;8(1):21-6.
- [Background] Cramer H, Lauche R, Haller H, Steckhan N, Michalsen A, Dobos G. Effects of yoga on cardiovascular disease risk factors: a systematic review and meta-analysis. Int J Cardiol. 2014 May 1;173(2):170-83. doi: 10.1016/j.ijcard.2014.02.017. Epub 2014 Feb 25. PMID 24636547
- [Background] Birdee GS, Ayala SG, Wallston KA. Cross-sectional analysis of health-related quality of life and elements of yoga practice. BMC Complement Altern Med. 2017 Jan 31;17(1):83. doi: 10.1186/s12906-017-1599-1. PMID 28143469
- [Background] Gordon L, McGrowder DA, Pena YT, Cabrera E, Lawrence-Wright M. Effect of exercise therapy on lipid parameters in patients with end-stage renal disease on hemodialysis. J Lab Physicians. 2012 Jan;4(1):17-23. doi: 10.4103/0974-2727.98665. PMID 22923917
- [Background] KauricKlein Z. Effect of yoga on physical and psychological outcomes in patients on chronic hemodialysis. Complement Ther Clin Pract. 2019 Feb;34:41-45. doi: 10.1016/j.ctcp.2018.11.004. Epub 2018 Nov 7. PMID 30712744
- [Background] Manaf, A. (2012). Yoga Asana The Art of Body Exercise (3. Baskı). İstanbul: Şan Ofset Baskı.
- [Background] Ünlü, B. (2007). Yoga For Everyone (B. Özükan, Ed.). İstanbul: Boyut Publishing.
- [Background] Krishna BH, Pal P, G K P, J B, E J, Y S, M G S, G S G. Effect of yoga therapy on heart rate, blood pressure and cardiac autonomic function in heart failure. J Clin Diagn Res. 2014 Jan;8(1):14-6. doi: 10.7860/JCDR/2014/7844.3983. Epub 2014 Jan 12. PMID 24596712
- [Background] Hartley L, Dyakova M, Holmes J, Clarke A, Lee MS, Ernst E, Rees K. Yoga for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2014 May 13;2014(5):CD010072. doi: 10.1002/14651858.CD010072.pub2. PMID 24825181
- [Background] Manchanda SC. Yoga--a promising technique to control cardiovascular disease. Indian Heart J. 2014 Sep-Oct;66(5):487-9. doi: 10.1016/j.ihj.2014.08.013. Epub 2014 Oct 8. No abstract available. PMID 25443600
- [Background] Jones SM, Guthrie KA, Reed SD, Landis CA, Sternfeld B, LaCroix AZ, Dunn A, Burr RL, Newton KM. A yoga & exercise randomized controlled trial for vasomotor symptoms: Effects on heart rate variability. Complement Ther Med. 2016 Jun;26:66-71. doi: 10.1016/j.ctim.2016.03.001. Epub 2016 Mar 4. PMID 27261984
- [Background] Wahlstrom M, Rydell Karlsson M, Medin J, Frykman V. Effects of yoga in patients with paroxysmal atrial fibrillation - a randomized controlled study. Eur J Cardiovasc Nurs. 2017 Jan;16(1):57-63. doi: 10.1177/1474515116637734. Epub 2016 Jul 7. PMID 26976659
- [Background] Barrows JL, Fleury J. Systematic Review of Yoga Interventions to Promote Cardiovascular Health in Older Adults. West J Nurs Res. 2016 Jun;38(6):753-81. doi: 10.1177/0193945915618610. Epub 2015 Dec 21. PMID 26689218
- [Background] Howie-Esquivel J, Lee J, Collier G, Mehling W, Fleischmann K. Yoga in heart failure patients: a pilot study. J Card Fail. 2010 Sep;16(9):742-9. doi: 10.1016/j.cardfail.2010.04.011. Epub 2010 Jun 8. PMID 20797598
- [Background] Taylor RS, Sagar VA, Davies EJ, Briscoe S, Coats AJ, Dalal H, Lough F, Rees K, Singh S. Exercise-based rehabilitation for heart failure. Cochrane Database Syst Rev. 2014 Apr 27;2014(4):CD003331. doi: 10.1002/14651858.CD003331.pub4. PMID 24771460
- [Background] Kuehn BM. Emerging Data Support Benefits of Yoga for Patients With Heart Disease. Circulation. 2017 Jan 24;135(4):398-399. doi: 10.1161/CIRCULATIONAHA.116.026989. No abstract available. PMID 28115415
- [Background] Hagglund E, Hagerman I, Dencker K, Stromberg A. Effects of yoga versus hydrotherapy training on health-related quality of life and exercise capacity in patients with heart failure: A randomized controlled study. Eur J Cardiovasc Nurs. 2017 Jun;16(5):381-389. doi: 10.1177/1474515117690297. Epub 2017 Jan 27. PMID 28128646
- [Background] Kwong JS, Lau HL, Yeung F, Chau PH. Yoga for secondary prevention of coronary heart disease. Cochrane Database Syst Rev. 2015 Jul 1;2015(7):CD009506. doi: 10.1002/14651858.CD009506.pub4. PMID 26130018
- [Background] Pullen PR, Thompson WR, Benardot D, Brandon LJ, Mehta PK, Rifai L, Vadnais DS, Parrott JM, Khan BV. Benefits of yoga for African American heart failure patients. Med Sci Sports Exerc. 2010 Apr;42(4):651-7. doi: 10.1249/MSS.0b013e3181bf24c4. PMID 19952833
- [Background] Guddeti RR, Dang G, Williams MA, Alla VM. Role of Yoga in Cardiac Disease and Rehabilitation. J Cardiopulm Rehabil Prev. 2019 May;39(3):146-152. doi: 10.1097/HCR.0000000000000372. PMID 31021995
- [Background] Akyol, A., Yesilbalkan, O. U., Kutlay, E., Kankaya, H., Menekli, T., & Fadiloglu, C. (2018). The Effects of Exercise on Quality of Life and Physiological Parameters in Obese Nursing Students/Obez Hemsirelik Ogrencilerinde Egzersizin Yasam Kalitesi ve Fizyolojik Parametrelere Olan Etkisi. Journal of Education and Research in Nursing, 15(3), 161-170.
- See also: World Health Organization (2021). Cardiovascular Diseases. Accessed on 26.07.2021 from https://www.who.int/health-topics/cardiovascular-diseases#tab=tab_1. — https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)?gad_source=1&gclid=EAIaIQobChMIo5Xp6t6lhQMVMZFoCR0iUg3rEAAYASAAEgKTp_D_BwE